CLINICAL TRIAL: NCT01139879
Title: Assessment of the Incidence and Treatment of Stage II -IV Pressure Ulcers in the Home Care or Extended Care Environments Utilizing the P400 Mattress
Brief Title: P400 for Stage II-IV Pressure Ulcers in Home and Extended Care
Acronym: P400
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hill-Rom (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-0092
Record Dates: First submitted 2010-06-07; First posted 2010-06-09 (Estimated); Results first posted 2015-12-17 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-11

CONDITIONS: Pressure Ulcers
Keywords: Pressure Ulcer treatment Mattresses; Home Care; Extended Care; Wound measurements
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- P400 support surface (Experimental): All patients will receive the P400 mattress
  Interventions: Device: P400 mattress

INTERVENTIONS:
Device: P400 mattress — The P400 mattress will be placed for a period of 12 weeks.

SUMMARY:
To assess the efficacy of a pressure ulcer treatment mattress, the P400 mattress, in the treatment of multiple Stage II or one or more large Stage III or IV pressure ulcers in the home care and extended care (nursing home) environment.

DETAILED DESCRIPTION:
Subjects will be recruited from those presenting to the wound clinic and meet the inclusion criteria. A total of 30 evaluable subjects will be recruited for this study from up to 2 wound care clinics /home health agencies (15 in Home Care and 15 in Extended Care). Subjects will be followed by weekly wound assessments for a period of 12 weeks or until their wounds heal. The outcome measurement is the rate of healing over the 12 week period.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has multiple Stage II pressure ulcers or at least one Stage III or IV pressure ulcer(s) (as per National Pressure Ulcer Advisory Panel Staging guidelines) located either on the trunk or pelvis (which would include trochanter and ischial ulcers ) having a clean wound bed of less than or equal to 25% necrotic tissue at the base of the pressure ulcer.
2. Subjects may have heel ulcers, however these ulcers may not be considered a target study ulcer.
3. Subject, or legally authorized representative is able to provide informed consent
4. Subject weighs between 70 and 350 pounds
5. Subject's nutritional status is thought to be adequate to support wound healing
6. Subject qualifies for a Group 2 support surface (Target study ulcer must be at least 8 cm^2 in area to qualify)

Exclusion Criteria:

1. Subject's target ulcer is unstageable due to eschar or necrosis or a suspected Deep Tissue Injury may be located at the base of the wound.
2. Subject has unresolved systemic infection, or pressure ulcer infection, or a history of osteomyelitis, or greater than 25% eschar or necrotic tissue present in the wound bed.
3. Patient has already been enrolled in this study
4. Patient has a recent history of non-compliance with pressure ulcer offloading, repositioning, or other areas of the treatment care plan, which would jeopardize wound healing if continued.
5. Care plan goals are palliative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall Wolcott, MD, Principal Investigator — Randall Wolcott and Assoiciates
Locations (1):
- Southwest Regional Wound Care Center, Lubbock, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- P400: All patients will receive the P400 mattress
  P400 mattress: The P400 mattress will be placed for a period of 12 weeks.
Period: Overall Study
Arm/Group | P400
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients with multiple Stage II or at least one Stage III or IV pressure ulcer having less than or equal to 25% necrotic tissue present in the pressure ulcer at the time of placement.
Arm/Group | P400
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (21.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Ulcer Surface Area at Week 12
Description: The primary outcome measure for this study is to be healing rate by area, based on the identified target study ulcer.
Time Frame: 12 Weeks
Population: Ulcers decreased an average of 7.96 cm^2 (+/- 8.1 cm^2) over the 12 week period
Measure: Mean (Standard Deviation); unit: cm^2
Units Other Than Participants: All Pressure Ulcers
Arm/Group | P400 Support Surface
Number analyzed (Participants) | 10
Number analyzed (All Pressure Ulcers) | 29
cm^2 | -7.96 (8.1)

2. Secondary Outcome: Incidence of New Ulcers
Description: incidence of new ulcers while on the study surface
Time Frame: 12 Weeks
Measure: Number; unit: percentage of participants
Groups:
- P400: The P400 mattress will be placed for a period of 12 weeks for all enrolled patients
Arm/Group | P400
Number analyzed (Participants) | 10
percentage of participants | 0

3. Secondary Outcome: Healing Rate Per Week
Description: The mean change in area per week for all ulcers
Time Frame: 12 weeks
Population: Rate of change in area (healing) for all ulcers on all subjects in area (cm^2)/week
Measure: Mean (Standard Deviation); unit: cm^2/week
Units Other Than Participants: all ulcers
Groups:
- P400 Support Surface: All patients will receive the P400 mattress for a period of 12 weeks
Arm/Group | P400 Support Surface
Number analyzed (Participants) | 10
Number analyzed (all ulcers) | 29
cm^2/week | -0.92 (.79)

ADVERSE EVENTS:
Arm/Group | P400 Support Surface
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
Small study with no comparative arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No